CLINICAL TRIAL: NCT03685864
Title: Suture Embedding Acupuncture for Chronic Low Back Pain: A Randomized, Sham-Controlled Clinical Trial
Brief Title: Suture Embedding Acupuncture for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Meng-Huang Wu, Attending physician, Department of Orthopedics, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201807035
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture Embedding Acupuncture (Experimental): Suture Embedding Acupuncture 1 time for two weeks, total 3 times.
  Interventions: Other: Suture Embedding Acupuncture
- Sham acupuncture (Sham Comparator): Sham Acupuncture 1 time for two weeks, total 3 times.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Suture Embedding Acupuncture — Suture Embedding Acupuncture at 8 acupoints (both sides of BL23, BL24, BL25, BL37). Receiving intervention 1 time in 2 weeks, and total receive 3 times.
  Arms: Suture Embedding Acupuncture
Other: Sham Acupuncture — Sham Acupuncture at 8 acupoints (both sides of BL23, BL24, BL25, BL37). Receiving intervention 1 time in 2 weeks, and total receive 3 times.
  Arms: Sham acupuncture

SUMMARY:
Chronic low back pain (cLBP) is a common public health issue, and it is one of the main causes of disability among adults of working age. Suture embedding acupuncture is one of the most often used interventions for the treatments of cLBP. The investigators will investigate the efficacy and safety of suture embedding acupuncture for cLBP in this single center, parallel, randomized, sham-controlled clinical trial.

DETAILED DESCRIPTION:
Suture embedding acupuncture is one of the most often used interventions for the treatments of chronic low back pain (cLBP). The investigators will investigate the efficacy and safety of suture embedding acupuncture for cLBP in this single center, parallel, randomized, sham-controlled clinical trial.

Participants will be randomized into 2 groups (real acupuncture and sham acupuncture) by central allocation. Randomized participants will complete a questionnaire that solicited information regarding age, sex, marital status, occupation, education, and medical history. The blinding credibility of the treatments will be evaluated at the end of the treatment.

Real Suture embedding Acupuncture for Treatment Group To make the real suture embedding acupuncture treatment reflect an ordinary clinical practice condition, participants received standardized acupuncture treatment. That treatment was accomplished by selecting a group of acupuncture points that predefined. Acupuncture points will be bladder meridian pattern acupuncture points including Shenshu (BL23), Qihaishu (BL24), Dachangshu (BL25), and Yimmen (BL37). Treatment will be given using sterile, disposable stainless steel 23G or 25G injection needles with 1 mm 5.0 Vicryl suture inside the needle. The needles will be inserted perpendicular to a depth of 5 to 35 mm depending on the acupuncture point, which was followed by manual stimulation by bidirectional rotation to induce Deqi sensation. Deqi was defined as a dull, localized, and aching sensation, which signaled the attainment of qi. After the Deqi sensation being achieved, the suture will be embedded with a sterile stainless steel needle. After needle removal, a 5mm × 5 mm sterile tape will be adhered to the needle hole. Patients will be asked not to remove the tape unless necessary.

Sham Acupuncture for Control Group Treatment will be given using sterile, disposable stainless steel 30G or 32G acupuncture needles. The acupuncture points will be the same as real suture embedding acupuncture group. The needles will be inserted perpendicular to a depth of 5 to 35 mm depending on the acupuncture point and will be pulled up immediately. After sham acupuncture, the point will be adhered a sterile tape as real group. Patients will be asked not to remove the tape unless necessary.

Outcome Measures Primary Outcome Measure The primary outcome measure is VAS for LBP. To understand the impact of cLBP on the participants' life, VAS for bothersomeness is chosen instead of pain intensity. The participants will be asked to mark, on a 10 cm VAS (0, absence of bothersomeness; 10, the worst bothersomeness imaginable), the average degree of bothersomeness due to LBP experienced within the most recent 1 week from the day of the assessment. This measurement has substantial validity. Bothersomeness of LBP will be measured at baseline, 2-, 4-, 8-, 12-, 16-, 20-, and 24-week. The primary endpoint is the 8-week follow-up (i.e., 4 wk after finishing all of the treatments).

Secondary Outcome Measures VAS for pain intensity is a simple method evaluating the subjective intensity of pain. Pain intensity will be measured in the same way as VAS for bothersomeness. Validity of its reliability has been demonstrated. The Chinese version Oswestry Disability Index (ODI) is used to measure back pain-related dysfunction. Health-related quality of life will be measured using the well-validated EuroQol 5 dimensions (EQ-5D). A higher score is indicative of a better general health status. Participants satisfaction will be evaluated with 5 point scale (1 is worst, and 5 is best)

Statistical Analyses To determine appropriate sample size, the VAS mean difference between the 2 groups will be assumed to be 1.5 and standard deviation to be 2.73 cm with significance level([alpha]) = 0.05 and power(1-ß) = 0.80. For the equal allocation for the 2 groups, total sample size considering dropout rate of 20% will be calculated as 130 subjects, which means that at least 104 subjects would finally be required after drop outs. The investigators performed the Shapiro-Wilk normality test to determine whether or not the sample values followed a normal distribution and finally assumed normality according to the test result. For all statistical analysis, SPSS 18.0 (SPSS Inc., Chicago, IL) will be used. Significance level will be set at P < 0.05. Per protocol (PP) analysis included all participants randomized and followed up until the last follow-up point.

ELIGIBILITY:
Inclusion Criteria:

* cLBP lasting for at least the last 3 months.
* 10-cm visual analogue scale (VAS) for bothersomeness of LBP exceeding 4.
* Nonspecific and uncomplicated LBP that was intact on neurological examination.

Exclusion Criteria:

* Exclusion criteria are sciatic pain (i.e., if a patient reported typical radiating pain in the leg as well as one or more neurological indications of nerve root tension or neurological deficit)
* Pain mainly below the knee; serious spinal disorders including malignancy, vertebral fracture, spinal infection, inflammatory spondylitis and cauda equine compression; history of previous spinal surgery or scheduled surgery to address a chronic disease that could interfere with treatment effects (e.g., cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, dementia, and epilepsy);
* Acupuncture treatment of LBP during the previous month
* Conditions that could compromise the safety of acupuncture (e.g., clotting disorders, taking anticoagulant agent, pregnancy, and seizure disorders);
* Severe psychiatric or psychological disorder
* Use of corticosteroids, narcotics or herbal medicine to treat LBP within one month.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
VAS | 2 week
  The patients will be asked to mark, on a 10 cm VAS (0, absence of bothersomeness; 10, the worst bothersomeness imaginable)

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 2 week
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel
EQ-5D | 2 week
  In description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  In evaluation part, the respondents evaluate their overall health status using the visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Huang Lin, PhD, Study Chair — Taipei Medical University
Locations (1):
- Taipei medical university hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan Z. Observation on 105 cases of duodenal bulbar ulcer treated by combined therapy of catgut embedding and Chinese drugs. J Tradit Chin Med. 2001 Jun;21(2):111-5. No abstract available. PMID 11498898
- [Background] Cho YJ, Song YK, Cha YY, Shin BC, Shin IH, Park HJ, Lee HS, Kim KW, Cho JH, Chung WS, Lee JH, Song MY. Acupuncture for chronic low back pain: a multicenter, randomized, patient-assessor blind, sham-controlled clinical trial. Spine (Phila Pa 1976). 2013 Apr 1;38(7):549-57. doi: 10.1097/BRS.0b013e318275e601. PMID 23026870
- [Background] Manheimer E, White A, Berman B, Forys K, Ernst E. Meta-analysis: acupuncture for low back pain. Ann Intern Med. 2005 Apr 19;142(8):651-63. doi: 10.7326/0003-4819-142-8-200504190-00014. PMID 15838072